CLINICAL TRIAL: NCT01529684
Title: A Phase 1, Open-label Study to Investigate the Absorption, Metabolism, and Excretion of 14C-OSI-906 in Subjects With Advanced Solid Tumors With an Optional Treatment Phase
Brief Title: A Study to Look at How a Single Oral Dose of 14C-OSI-906 is Absorbed, Broken Down and Eliminated in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OSI-906-104
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors; Pharmacokinetics of 14C-OSI-906
Keywords: oncology patients; Metabolic profile of 906; OSI-906; mass balance; Pharmacokinetics of 14C-OSI-906; Cancer, solid tumors; Absorption, Metabolism, and Excretion of OSI-906
MeSH Terms: conditions — Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OSI-906 (Experimental): Two Parts:
  Part A: 14C-labeled OSI-906
  Part B: (Optional) OSI-906 (non-labeled)
  Interventions: Drug: radio-labeled OSI-906; Drug: OSI-906

INTERVENTIONS:
Drug: radio-labeled OSI-906 — Part A: oral solution of 14C-OSI-906
Drug: OSI-906 — Part B: oral tablets OSI-906

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, in particular the routes of excretion and extent of metabolism of OSI-906 after a single oral dose of 14C-labeled OSI-906. Subjects with Advanced Solid Tumors may participate and then continue into the Optional Treatment Phase.

DETAILED DESCRIPTION:
This study includes two parts: Part A

Subjects will be admitted to the clinical research unit on Day -1 and remain confined to the unit until post dosing discharge criteria are met up to a maximum of 10 days. On Day 1, subjects will receive a single oral dose of 14C-labeled OSI-906.

Part B (optional)

Once the subject has completed part A, the subject may elect to continue participation in Part B. Subjects will receive OSI-906 (non-radiolabeled) twice daily by mouth. Subjects will be seen for scheduled visits every 7 days for the first 36 days and then every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histologically or cytologically confirmed diagnosis of advanced solid tumor (measurable or non-measurable disease) for which no conventional therapy is available
* The subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
* The subject has a predicted life expectancy ≥12 weeks
* The subject has a fasting glucose ≤125 mg/dL (7 mmol/L) at Screening, Day -1 and pre-dose Day 1
* The subject has adequate organ function defined by the following laboratory parameters:

  * absolute neutrophil count (ANC) ≥1.5 x 10 9/L
  * platelet count ≥100 x 10 9/L
  * total bilirubin ≤1.5 x upper limit of normal (ULN)
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN if subject has documented liver metastases
  * serum creatinine ≤1.5 x ULN
  * potassium, calcium, and magnesium within normal limits or determined by the investigator to be not clinically significant (NCS)
* The subject has a negative cotinine test
* If male, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method while participating in the study and for 90 days after the last dose of study medication
* If female, the subject is surgically sterile or status post hysterectomy, post-menopausal, or is using 2 forms of medically acceptable methods of birth control, one of which must be a barrier method to prevent pregnancy and agrees to continue using this method from screening until 90 days after the last dose of study medication
* If female, the subject must not be breastfeeding at Screening, during the study period and for 90 days after last dose of study drug administration
* If female, the subject must not donate ova starting at Screening, and throughout the study period and for 90 days after last dose of study drug administration
* Female subject of child bearing potential has a negative pregnancy test at Screening and Day -1

Exclusion Criteria:

* The subject has Type 1 or Type 2 diabetes mellitus currently requiring insulinotropic or insulin therapy
* The subject has a history of poorly controlled gastrointestinal disorder (s) that could affect the absorption or metabolism of study drug
* The subject has used IGF-1R inhibitor therapy in last 6 months
* The subject has hepatocellular carcinoma
* The subject has used a CYP1A2 inhibitor or inducer within 14 days prior to Day 1
* The subject has used drugs with a risk of causing QTc interval prolongation and Torsade de Pointes (TdP) within 14 days prior to Day 1
* The subject has a history (within last 6 months) of significant cardio-vascular disease
* The subject has a history (within the last 6 months) of significant arrhythmia disease, unless the disease is well-controlled with medication per the Principal Investigator's clinical judgment
* The subject has had major surgery ≤ 3 weeks prior to Day 1
* The subject has had radiation ≤ 3 weeks prior to Day 1
* The subject has had chemotherapy ≤ 3 weeks prior to Day 1
* The subject has participated in a radiolabeled study in the last 12 months
* The subject has a history of cerebrovascular accident (CVA) within 6 months prior to Day 1 or that resulted in ongoing neurologic instability
* The subject has an active infection or serious underlying medical condition (including any type of active seizure disorder within 12 months prior to Day 1) that would impair the ability of the subject to receive study drug
* The subject has participated in any interventional clinical study within 21 days or has been treated with any investigational drugs within 30 days or 5 half lives whichever is longer, prior to the initiation of Screening
* The subject has a history of any psychiatric condition that might impair the subject's ability to understand or to comply with the requirements of the study or to provide informed consent
* The subject is pregnant or lactating
* The subject has symptomatic brain metastases that are not stable, require steroids, or that have required radiation and/or other related treatment, (i.e., anti-epileptic medication) within 28 days prior to Day 1
* The subject has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03-19 (Actual); Primary Completion 2012-12-08 (Actual); Study Completion 2013-02-20 (Actual)

PRIMARY OUTCOMES:
Radioactivity in whole blood and plasma | Up to 10 days from time of receipt of 14C-labeled OSI-906
  Outcome measure for Part A: Area under the time concentration curve extrapolated to infinity (AUCinf), AUC from time of dosing to last quantifiable time point (AUClast), Maximum Plasma Concentration (Cmax), Time to maximum concentration (Tmax), Terminal half-life (t 1/2), Apparent Body Clearance after dosing (CL/F), and Apparent volume of distribution (Vz/F)
Radioactivity ratio in blood/plasma | Up to 10 days from time of receipt of 14C-labeled OSI-906
  Outcome Measure for Part A of OSI-906 distribution between cellular components and plasma
Excretion ratio and cumulative excretion of radioactivity in urine and feces | Up to 10 days from time of receipt of 14C-labeled OSI-906
  Outcome measure for Part A
Composite of Pharmacokinetics of OSI-906 in plasma: AUC inf, AUC last, C max, t max, t 1/2, CL/F, and Vz/F | Up to 10 days from time of receipt of 14C-labeled OSI-906
  Outcome measure for Part A
Composite of Pharmacokinetics of OSI-906 in urine: Cumulative amount of drug excreted into urine, feces or bile up to collection time of last measurable concentration (Ae last), Renal Clearance (CL R), and percentage of dose excreted (Ae last%) | Up to 10 days from time of receipt of 14C-labeled OSI-906
  Outcome measure for Part A

SECONDARY OUTCOMES:
Metabolic Profile: Profiling of possible metabolites in OSI-906 plasma, urine, and feces | Up to 10 days from time of receipt of 14C-labeled OSI-906
  Outcome measure for Part A
Safety as assessed by recording adverse events, laboratory assessments and vital signs, and electrocardiograms (ECGs) | For Part A: Days 1-10 and/or 30 days post treatment visit. For Part B: Treatment Period 1 (TP1) through 30 day post treatment visit (up to two years)
  Outcome measures for Part A and Part B

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (2):
- United States (2):
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Comprehensive Clinical Development NW, Inc., Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=269